CLINICAL TRIAL: NCT01213966
Title: Phase IIa Exploratory, Open Label, Single/Multiple Dose Testing Clinical Study to Assess the Preliminary Efficacy, Tolerability and PK of OZ439 in Adult Patients With Acute, Uncomplicated P. Falciparum or Vivax Malaria Mono-infection
Brief Title: Efficacy, Tolerability, PK of OZ439 in Adults With Acute, Uncomplicated P.Falciparum or Vivax Malaria Mono-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMV_OZ439_10_002
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Malaria, Falciparum; Malaria, Vivax
Keywords: Acute uncomplicated Plasmodium Falciparum malaria; Blood stage Plasmodium Vivax malaria
MeSH Terms: conditions — Malaria, Falciparum; Malaria, Vivax | interventions — artefenomel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 800 mg OZ439 po single dose (Experimental): 800 mg OZ439 po single dose
  Interventions: Drug: OZ439
- 400 mg OZ439 p.o. single dose (Experimental): 400 mg OZ439 p.o. single dose
  Interventions: Drug: OZ439
- 200mg OZ439 p.o. single dose (Experimental): 200mg OZ439 p.o. single dose
  Interventions: Drug: OZ439
- 1200 mg OZ439 po single dose (Experimental): 1200 mg OZ439 po single dose
  Interventions: Drug: OZ439

INTERVENTIONS:
Drug: OZ439 — po, single dose
  Other Names: Artefenomel

SUMMARY:
A Phase IIa Exploratory, Open label, Single Dose Regimen, Multiple Dose Testing Clinical Study to Assess the Preliminary Efficacy, Tolerability and Pharmacokinetics of OZ439 in adult patients with acute, uncomplicated Plasmodium falciparum or vivax malaria mono-infection.

DETAILED DESCRIPTION:
This exploratory Phase IIa study aims to investigate the preliminary efficacy in terms of parasite reduction and clearance in malaria patients, and the tolerability of OZ439 administered as single dose regimen at 3 different doses in parallel cohorts of patients with either acute uncomplicated Plasmodium falciparum or Plasmodium vivax malaria mono-infection (10 patients per plasmodium species per dose level).

Treatment with OZ439 will be given as a single dose on Day 0, starting in the first cohort at a dose of 800 mg. Established antimalarial therapy will be given at the latest at 36 hours post dosing.

The primary endpoint will be the derived parasite reduction rate (PRR) at 24 hours after study drug administration.

A review of each individual study cohort (dose/species) will be conducted with the Principal Investigator and the Sponsor and a decision will be reached on whether the dose for the next cohort should increase or decrease (within 200mg-1600mg range). This decision will be based on parasite reduction rate over the first 24 hours following administration of OZ439, tolerability and exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the age of 18 and 60 years, inclusive
2. Body weight between 40 kg and 90 kg inclusive
3. Presence of mono-infection of P. falciparum or P. vivax confirmed by:

   * Fever, as defined by axillary temperature ≥ 37.5°C or oral/rectal/tympanic temperature ≥ 38°C, or history of fever in the previous 24 hours (history of fever must be documented) and,
   * Microscopically confirmed parasite infection, 5,000 to 50,000 asexual parasite count/µl of blood
4. Written informed consent, in accordance with local practice, provided by patient. If the patient is unable to write, witnessed consent is permitted according to local ethical considerations
5. Ability to swallow oral medication
6. Ability and willingness to participate and access the health facility
7. Agree to minimum of 4 days hospitalisation for drug administration and pharmacokinetic sampling

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria requiring parenteral treatment according to the World Health Organisation Criteria 2010 (Attachment 2)
2. Mixed Plasmodium infection
3. Severe vomiting, defined as more than three times in the 24 hours prior to inclusion in the study or inability to tolerate oral treatment, or severe diarrhoea defined as 3 or more watery stools per day
4. Presence of other serious or chronic clinical condition requiring hospitalisation.
5. Severe malnutrition (defined as the weight-for-height being below -3 standard deviation or less than 70% of median of the NCHS/WHO normalised reference values).
6. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, QTc interval greater than or equal to 450 msec), respiratory (including active tuberculosis), history of jaundice, hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric, history of convulsions or other abnormality (including head trauma).
7. Known history of hypersensitivity, allergic or adverse reactions to artemisinin containing compounds or mefloquine or drug in the national guidelines for P. vivax.
8. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab).
9. Have received any antimalarial treatment in the preceding 14 days, as determined by history and screening test.
10. Have received antibacterial with known antimalarial activity in the preceding 14 days.
11. Have received an investigational drug within the past 4 weeks.
12. Liver function tests (ASAT/ALAT levels) more than 2 x ULN
13. Hb level below 10 g/dL.
14. Bilirubin levels greater than 40 µmol/L.
15. Serum creatinine levels more than 2 times the upper limit of normal range in absence of dehydration. In case of important dehydration the creatinine should be lower than 2X ULN after oral/parenteral rehydration.
16. Female patients must be neither pregnant (as demonstrated by a negative serum pregnancy test) nor lactating, and must be willing to take measures not to become pregnant during the study period and safety follow-up period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2010-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sasithon Pukrittayakamee, MD, Principal Investigator — Mahidol University

REFERENCES:
- [Derived] Phyo AP, Jittamala P, Nosten FH, Pukrittayakamee S, Imwong M, White NJ, Duparc S, Macintyre F, Baker M, Mohrle JJ. Antimalarial activity of artefenomel (OZ439), a novel synthetic antimalarial endoperoxide, in patients with Plasmodium falciparum and Plasmodium vivax malaria: an open-label phase 2 trial. Lancet Infect Dis. 2016 Jan;16(1):61-69. doi: 10.1016/S1473-3099(15)00320-5. Epub 2015 Oct 5. PMID 26448141

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at two study centres in Thailand Primary study centre: Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand Sub-centre: Shoklo Malaria Research Unit, Mae Sod, Tak, Thailand The first patient was enrolled on 24 October 2010 and the last patient completed on 25 May 2012.
Pre-assignment Details: There was no washout, run-in or transition following enrolment but prior to group assignment.
Groups:
- 800 mg OZ439 po Single Dose: Cohort 1 received a dose of 800 mg. The decision to decrease and/or increase the dose (within a 100 mg to 1600 mg range) in each next cohort of patients was made following a study cohort review
- 400 mg OZ439 p.o. Single Dose; 200mg OZ439 p.o. Single Dose: Ultimately, after review of the data from Cohort 1 (800 mg), patients in Cohort 2 received 400 mg OZ439, patients in Cohort 3 received 200 mg OZ439, and patients in Cohort 4 received 1200 mg OZ439.
- 1200 mg OZ439 po Single Dose: Ultimately, after review of the data from Cohort 1 (800 mg), patients in Cohort 2 received 400 mg OZ439, patients in Cohort 3 received 200 mg OZ439, and patients in Cohort 4 received 1200 mg OZ439.received single dose
Period: Overall Study
Arm/Group | 800 mg OZ439 po Single Dose | 400 mg OZ439 p.o. Single Dose | 200mg OZ439 p.o. Single Dose | 1200 mg OZ439 po Single Dose
Started | 20 | 20 | 20 | 21
Completed | 19 | 20 | 17 | 20
Not Completed | 1 | 0 | 3 | 1
Not completed — Protocol Violation | 1 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - OZ439 800mg: 800 mg OZ439 po single dose
- Cohort 2 - OZ439 400mg: 400 mg OZ439 p.o. single dose
- Cohort 3 - OZ439 200mg: 200mg OZ439 p.o. single dose
- Cohort 4 - OZ439 1200mg: 1200 mg OZ439 po single dose
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - OZ439 800mg | Cohort 2 - OZ439 400mg | Cohort 3 - OZ439 200mg | Cohort 4 - OZ439 1200mg | Total
Number analyzed (Participants) | 20 | 21 | 20 | 21 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 20 | 21 | 82
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (8.37) | 29.1 (9.82) | 26.7 (9.75) | 29.3 (8.19) | 28.1 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 4 | 11
  Male | 18 | 17 | 19 | 17 | 71
Region of Enrollment [Number; unit: participants]
  Thailand | 20 | 21 | 20 | 21 | 82

OUTCOME MEASURES:

1. Primary Outcome: Derived Parasite Reduction Rate at 24 Hours (PPR24)
Description: PRR24 is the log10 change in parasitemia over 24 hours estimated from a regression model fit separately for each patient. The relationship between parasite counts and time was analyzed by fitting a variable lag phase, then a linear decline to the natural log of parasite count versus time relationship. The slope of this log linear relationship is the primary end-point.
  The time points chosen for the regression are those that yield the highest degree of significance when assessing the regression when the number of time points are greater than or equal to 3. No extrapolation was performed.
Time Frame: 24 hours after study drug administration
Measure: Median (Full Range); unit: Log10 parasites/24h
Groups:
- 800 mg OZ439 po Single Dose: The first cohort received a dose of 800 mg. The decision to decrease and/or increase the dose (within a 100 mg to 1600 mg range) in each next cohort of patients with either P. falciparum or P. vivax malaria, was made following a study cohort review of the safety data, drug exposure levels, and the PRR over 24 hours after the investigational product administration (PRR24) obtained from the previous cohort.
- 400 mg OZ439 p.o. Single Dose: After review of the data from Cohort 1 (800 mg), patients in Cohort 2 received a single dose of 400 mg OZ439.
- 200mg OZ439 p.o. Single Dose: Ultimately, after review of the data from Cohort 1 (800 mg) and data from Cohort 2 (400 mg), patients in Cohort 3 received a single dose of 200 mg OZ439.
- 1200 mg OZ439 po Single Dose: Ultimately, after review of the data from Cohort 1 (800 mg), from Cohort 2 (400 mg), and Cohort 3 (200 mg), patients in Cohort 4 received a single dose of 1200 mg OZ439.
  It was decided not to proceed with a fifth cohort and no further patients were enrolled.
Arm/Group | 800 mg OZ439 po Single Dose | 400 mg OZ439 p.o. Single Dose | 200mg OZ439 p.o. Single Dose | 1200 mg OZ439 po Single Dose
Number analyzed (Participants) | 19 | 20 | 17 | 20
Log10 parasites/24h
  PPR24 Plasmodium Falciparum | 1.38 [0.62 to 2.79] | 1.56 [1.29 to 3.11] | 1.71 [-1.69 to 1.88] | 1.63 [1.13 to 3.58]
  PPR24 Plasmodium Vivax | 2.05 [1.46 to 2.79] | 2.18 [0.99 to 3.59] | 2.40 [1.74 to 3.59] | 1.96 [1.86 to 3.09]
Statistical Analysis 1: Comparison: 800 mg OZ439 po Single Dose vs 400 mg OZ439 p.o. Single Dose vs 200mg OZ439 p.o. Single Dose vs 1200 mg OZ439 po Single Dose; PPR24 was summarised descriptively. No statistical test was performed; Test type: Superiority or Other; p = 0.01, Regression, Linear — PPR24 was summarized descriptively. No statistical test was performed. The PRR24 values were summarised when the corresponding regression fit had a p-value of p ≤0.01 and an adjusted coefficient of determination (R2) ≥0.85

ADVERSE EVENTS:
Time Frame: Adverse events reported from pre-dose to end of study visit. An SAE was to be monitored until resolution. Patients experiencing AEs were monitored for up to 30 days after the end of the study or resolution of the event, whichever was the earlier.
Arm/Group | Cohort 1 - OZ439 800mg | Cohort 2 - OZ439 400mg | Cohort 3 - OZ439 200mg | Cohort 4 - OZ439 1200mg
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 1/20 | 1/21
Other Adverse Events (participants affected / at risk) | 4/20 | 6/20 | 10/20 | 8/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - OZ439 800mg (N=20) | Cohort 2 - OZ439 400mg (N=20) | Cohort 3 - OZ439 200mg (N=20) | Cohort 4 - OZ439 1200mg (N=21)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — moderate, considered unrelated to the investigational product
Malaria relapse (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — moderate, considered not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - OZ439 800mg (N=20) | Cohort 2 - OZ439 400mg (N=20) | Cohort 3 - OZ439 200mg (N=20) | Cohort 4 - OZ439 1200mg (N=21)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Creatine PK Increased (Investigations) | 1 (1) | 1 (1) | 5 (5) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
ALAT Increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
ASAT Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ECG QT Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECG T Wave Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heamoglobin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less